CLINICAL TRIAL: NCT01635855
Title: Belotero® Post Approval Study for the Treatment of Nasolabial Folds
Brief Title: Belotero Post Approval Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110637
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belotero (Experimental): Belotero® Hyaluronic acid dermal filler
  Interventions: Device: Belotero®

INTERVENTIONS:
Device: Belotero® — Hyaluronic acid dermal filler

SUMMARY:
A prospective, open-label 1-month post-approval study to evaluate the short term safety of Belotero® Balance in the re-treatment of nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

1. Was a participant in the Belotero® Balance pre-market IDE clinical trial or the Belotero Balance Fitzpatrick Skin Type IV-VI Study.
2. Is a candidate for bilateral nasolabial fold re-treatment with Belotero® Balance.
3. Understands and accepts the obligation not to receive any other facial procedures from enrollment through 1 month from optimal correction in the current study.
4. Understands and accepts the obligation to comply with the required follow-up visits and is logistically able to meet all study requirements.

Exclusion Criteria:

1. Has received surgery in either nasolabial fold.
2. Has received within the past 6 months a non-permanent filler (e.g. hyaluronic acid, CaHA) or neurotoxin below the zygomatic arch.
3. Has received at any time a permanent filler (e.g. polylactic acid, PMMA, silicone) below the zygomatic arch.
4. Has received within the past 6 months dermal resurfacing procedures (e.g. medium/deep chemical peel, dermabrasion treatments, ablative laser resurfacing) or non-invasive skin-tightening (e.g. Thermage) below the zygomatic arch.
5. Has received in the past 2 weeks prescription facial wrinkle therapies (e.g., RENOVA®), topical steroids, skin irritating topical preparations, or pigmenting agents (self-tanning agents) below the zygomatic arch.
6. Has received in the past 2 months or plans to receive during the study immunosuppressive medications or systemic steroids (intranasal / inhaled steroids acceptable).
7. Has an acute inflammatory process or infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events.
8. Has a known bleeding disorder or is using medication that reduces blood coagulation, (e.g. aspirin, non-steroidal anti-inflammatory drugs, or warfarin) which may increase the risk of bleeding during the treatment session.
9. Has a known history of severe allergies manifested by a history of anaphylaxis; or history or presence of multiple severe allergies.
10. Has known allergy or hypersensitivity to hyaluronic acid preparations, gram positive bacterial proteins or Belotero® or Belotero® derivative.
11. Has a known history of hyper- or hypo-pigmentation in the nasolabial folds, keloid formation, or hypertrophic scarring.
12. Is a female of childbearing potential (e.g. not post-menopausal for at least one year or has not had a hysterectomy or tubal ligation) and is pregnant, lactating or plans to become pregnant during the study or is not using medically effective birth control.
13. Has any other medical condition with the potential to interfere with the study or increase the risk of adverse events.
14. Is enrolled or plans to enroll in a competitive or interfering study.
15. Is an employee or direct relative of an employee of the investigational site or study sponsor.
16. All Fitzpatrick skin types are eligible for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Francisco, California
  - New Haven, Connecticut
  - Metairie, Louisiana
  - Glenn Dale, Maryland
  - Montclair, New Jersey
  - White Plains, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Belotero®: Hyaluronic Acid Dermal Filler: Belotero®: Hyaluronic acid dermal filler
Period: Overall Study
Arm/Group | Belotero®: Hyaluronic Acid Dermal Filler
Started | 117
Completed | 113
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The number of participants included in the analysis was per protocol. There were no imputation techniques used in the safety study.
Arm/Group | Belotero®: Hyaluronic Acid Dermal Filler
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.04 (9.40)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 117

OUTCOME MEASURES:

1. Primary Outcome: Rate of Severe Common Adverse Events
Description: The purpose of this study was to determine if the rate of "Severe" common adverse events after re-treatment with Belotero Balance differs from the combined rates reported in the Belotero® Balance IDE clinical trial and Belotero® Balance Fitzpatrick Skin Type IV-VI Study (Pre-Approval Studies)."Common" is defined as pre-specified adverse events occurring in >= 5% of study subjects. These averse events are: bruising, itching, pain, redness, swelling, discoloration, nodule, and induration.
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of 'severe' common AEs
Arm/Group | Belotero
Number analyzed (Participants) | 117
percentage of 'severe' common AEs | 8.5 [3.5 to 13.6]
Statistical Analysis 1: Comparison: Belotero; The analysis was performed by comparing the proportion of subjects with severe common adverse events in the post-market study to that occurred in the pre-market studies. It was pre-specified in the protocol that the proportion of subjects with severe common adverse events in the pre-market studies was 22%; Test type: Superiority or Other; p < 0.025, One sided binomial distribution — Ho (null): Ps >= 22% versus Ha (alternate): Ps < 22% where Ps is the proportion of subjects with common severe adverse events in the post-approval study. Ho is rejected if upper limit of the 95% CI of Ps < 22% and the one-sided p-value <= 0.025; The upper limit of the 95% two-sided CI for a proportion is equivalent to the 97.5% one-sided CI for that proportion for normal approximations; One-sided binomial = 8.5, 95% CI 2-sided [3.5 to 13.6]

ADVERSE EVENTS:
Time Frame: The purpose of this study was to determine the rate of "Severe" common adverse events after re-treatment with Belotero Balance differs from the combined rates reported in Belotero Balance IDE and Belotero Balance Fitzpatrick Skin Type IV-VI Study.
Arm/Group | Belotero®: Hyaluronic Acid Dermal Filler
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 100/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belotero®: Hyaluronic Acid Dermal Filler (N=117)
Bruising (Skin and subcutaneous tissue disorders) | 78
Itching (Skin and subcutaneous tissue disorders) | 31
Pain (Skin and subcutaneous tissue disorders) | 44
Redness (Skin and subcutaneous tissue disorders) | 68
Swelling (Skin and subcutaneous tissue disorders) | 79
Discoloration (Skin and subcutaneous tissue disorders) | 46
Nodule (Skin and subcutaneous tissue disorders) | 40
Induration (Skin and subcutaneous tissue disorders) | 19
Needle Jam (Investigations) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No manuscripts may be submitted for publication without prior review by the Sponsor. Investigator agrees to accommodate requests by Sponsor to protect proprietary rights/interests. Sponsor will be given full credit/acknowledgment for support provided for any publication resulting from this research. Investigator shall grant to the Sponsor an irrevocable royalty free, non-exclusive right to reproduce, translate, use all such copyrighted material arising from publications from study.